CLINICAL TRIAL: NCT05176613
Title: Effects of High Frequency Repetitive Transcranial Magnetic Stimulation Combined Motor Learning on Motor Function and Grip Force for Upper Limbs and Activities of Daily Living in Sub-acute Stroke Patients
Brief Title: Effects of High Frequency rTMS Combined Motor Learning on Upper Limb Motor Function in Subacute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chungnam National University Sejong Hospital (Other)
Responsible Party: Principal Investigator, JungWoo Shim, Principal Investigator, Chungnam National University Sejong Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016071HR
Record Dates: First submitted 2021-12-02; First posted 2022-01-04 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Stroke, Acute; Hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HF-rTMS and ML (Experimental): High frequency Repetitive Transcranial Magnetic Stimulation and Motor Learning(Experimental group)
  Interventions: Device: HF-rTMS; Behavioral: ML
- Sham-rTMS and ML (Sham Comparator): Sham Repetitive Transcranial Magnetic Stimulation and Motor Learning
  Interventions: Behavioral: ML; Device: Sham-rTMS

INTERVENTIONS:
Device: HF-rTMS — HF-rTMS stimulated a 70-mm, 8-shaped coil stimulator (The Magstim Company, UK, 2012) on the damaged cerebral cortex. Prior to the application of HF-rTMS, the motor point was identified that stimulates maximum thresholds on the primary motor cortex, causing flexion of the opposite index finger. If the cerebral hemisphere does not show a kinetic response even at the maximum stimulus, the motor point of the opposite hemisphere was found to be symmetrically changed. The intensity of the stimulus was 80% of the resting motor threshold, which means the motor eveked potential above which the first dorsal interosseous muscle can produce 50 μV more than five times out of 10 stimuli. The subject sat on a chair made to hold the head. The stimulation was stimulated at high frequency (10 Hz) for 2 seconds, and the rest was performed for 58 seconds for a total of 200 times for 10 minutes.
  Other Names: High Frequency repetitive Transcranial Magnetic Stimulation(HF-rTMS)
  Arms: HF-rTMS and ML
Behavioral: ML — Motor learning was conducted for two minutes each in five sessions, and the first is the external rotation training to maximum range of the shoulder joint in sitting position. The second method is to stack cups by transferring them from the non-affected side to the affected side by transferring 25 plastic cups of five colors in sitting position with both hands inserted. Third, by pushing and pulling the ball forward and backward with the hands folded, the subject puts a 55 cm healing ball on the table in a sitting position, and pushes and pulls it forward with the upper limb. The fourth method is to insert and remove pegs from the peg board, and the target uses the affected side hand in sitting position. The fifth method is to tear a newspaper, in which the subject overlaps a newspaper on the table in a sitting position, holds it with the non-affected hand, and tears it with the hands of the damage. A total of 10 minutes of motor learning.
  Other Names: Motor Learning(ML)
Device: Sham-rTMS — Sham rTMS gives a small intensity of 2% of the resting motor threshold that cannot cause excitement in the motor cortex, and is set to listen to the same frequency of noise as HF-rTMS, and motor learning is applied equally. A total of 20 minutes were applied three times a week for four weeks by applying 10 minutes of Sham rTMS and 10 minutes of motor learning.
  Other Names: Sham repetitive Transcranial Magnetic Stimulation(Sham-rTMS)
  Arms: Sham-rTMS and ML

SUMMARY:
This study is to present the effect of a program combining high frequency repetitive transcranial magnetic stimulation with motor learning on upper limb motor function and grip strength and activities of daily motion in patients with subacute stroke.

Purpose : This study was to investigate the effects of high frequency repetitive transcranial magnetic stimulation combined with motor learning effects motor function and grip force for upper limbs and activities of daily living of subacute stroke patients.

Subjects : Thirty individuals with subacute stroke, satisfying the selection criteria, were selected for this study. Subject were randomly allocated into 14 high frequency repetitive transcarnial magnetic stimulation+motor learning group(experimental group), 16 sham repetitive transcranial magnetic stimulation+motor learning group(control group).

Intervention : 12 sessions, 3d/wk, 4week Studies : upper limb functional assessment(FMA-U/L, BBT), hand grip force assessment(disital hand dynamometer), activities daily of living assessment(K-MBI) Evaluation : 1)pre test 2)post test

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegia from stroke
* Factors within six months of onset
* Found to have subcortex damage through diagnoses of magnetic resonance imaging(MRI)
* Had motor defects on the damaged upper extremities
* Korean version Mini mental state examination(MMSE-K) score greater than 24 points

Exclusion Criteria:

* Permanent damage such as heart vein
* Upper limb fractures
* Neurological damage such as Parkinson's, multiple sclerosis
* Other reasons limiting upper limb movement
* Epilepsy or family history of epilepsy
* wearing a metal tube in skull or pacemaker
* The lesion at occipital lobe

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05-13 (Actual); Primary Completion 2016-07-29 (Actual); Study Completion 2016-08-05 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer Assessment - Upper Limb(FMA-U/L) | Change from baseline at the end of four weeks intervention
  The FMA-U/L score is a tool for evaluating the body's structure, function, and activity level as an evaluation tool for evaluating motor function according to Brunnstrom's recovery phase of Step 6. The minimum value is 0 point and the maximum value is 66 points, and the higher the score, the better the outcome.

SECONDARY OUTCOMES:
Box and Block Test(BBT) | Change from baseline at the end of four weeks intervention
  The Box and Block Test(BBT) is device to assess upper limb dexterity in stroke patients
Digital hand dynamometer | Change from baseline at the end of four weeks intervention
  The digital hand dynamometer is device to assess hand grip force in stroke patients
Korean version of the Modified Barthel Index(K-MBI) | Change from baseline at the end of four weeks intervention
  The Korean version of the Modified Barthel Index (K-MBI) is a functional change sensitive evaluation tool. The minimum value is 0 point and the maximum value is 100 points, and the higher the score, the better the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: JungWoo Shim, master, Principal Investigator — Chungnam National University Hospital

IPD SHARING:
Plan to Share IPD: No